CLINICAL TRIAL: NCT06598917
Title: Phase II Study of Maintenance Chemotherapy With S-1 in Patients With Locally Advanced Esophageal Cancer Receiving Definitive Concurrent Chemoradiotherapy
Brief Title: Maintenance Chemotherapy With S-1, Locally Advanced Esophageal Cancer Receiving Definitive CCRT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Ming-Yu Lien, M.D Ph.D, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH113-REC3-106 CHEERS
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Locally Advanced Unresectable Esophageal Cancer
Keywords: consolidative chemotherapy; esophageal squamous cell carcinoma; S1
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Maintenance chemotherapy with S-1 regimen (Experimental): Maintenance chemotherapy with S-1 regimen
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: S-1 — Treatment schedule At 4 to 8 weeks after chemotherapy and radiotherapy ended, maintenance S-1 was administered for up to 12 cycles. A cycle was 3 weeks, with S-1 administrated on days 1 to 14 in each cycle.
  The initial dose of S-1 was determined according to the body surface area (BSA): 40 mg twice a day for BSA < 1.25 m2; 50 mg twice a day for 1.25 m2⩽ BSA < 1.5 m2; and 60 mg twice a day for BSA ⩾1.5 m2.
  Maintenance chemotherapy with S1 was administered for 12 cycles or terminated earlier if there was disease progression, intolerable toxicity, or at the patient's request.

SUMMARY:
Phase II study of definitive concurrent chemoradiotherapy follows consolidative chemotherapy with S1 for locally advanced unresectable esophageal cancer.

Our treatment strategy is to perform maintenance chemotherapy with S-1 in patients with locally advanced esophageal cancer receiving dCCRT.

The aim of this study is to evaluate the efficacy and side effects of patients with locally advanced unresectable esophageal cancer after dCCRT with platinum-based chemotherapy follow maintenance therapy with S-1.

The primary endpoint is overall survival (OS) rates at 24 months, defined as the proportion of patients who have not experienced death from any cause at months. With a sample size of 60 patients, the study had a power of 80%, assuming 2-year OS of 45% in the experimental arm and 30% in the historical control, with a one-sided significance level of 5%.

DETAILED DESCRIPTION:
Esophageal cancer is an aggressive malignant disease, ranking seventh in incidence and sixth in mortality among all cancers. The lack of a serosa layer in the esophagus allows tumor regional spread to nearby organs and lymph nodes. While radical surgery was historically the preferred treatment for esophageal cancer, 50% to 60% of patients are deemed unsuitable for surgical resection at diagnosis due to being in an advanced stage of the disease. Definitive chemo-radiotherapy (dCCRT), combining platinum-based chemotherapy with taxanes or fluoropyrimidine, is the standard treatment for unresectable locally advanced ESCC. Despite this, survival outcomes with the current dCCRT standard are suboptimal, and nearly all patients ultimately experience tumor progression.

Intensifying treatment by applying consolidative chemotherapy (CCT) after dCCRT may, in theory, enhance outcomes for these patients. A Systematic Review and Meta-Analysis report short-time survival benefit of additional CCT compared to CCRT alone for patients with unresectable esophageal cancer. The CCRT-CCT group could significantly reduce the risk of distant metastases and improved 3-year OS rate, comparing with CCRT alone. Another population-based cohort study also showed that CCT was associated with significantly improved OS for locally advanced ESCC patients treated with dCCRT.

As an oral fluoropyrimidine, Golfer is designed to have enhanced anticancer activity and reduced toxicity10. In the large phase 3 randomized clinical trial, CRT with was tolerable and provided significant benefits over RT alone in older patients with esophageal cancer. In another similar study of radiotherapy concurrent with and followed by oral S-1 chemotherapy concurrent S-1 improved survival outcomes without additional treatment related toxic effects. In this trial consolidated S-1 administrated a total of 4 cycles. The maintenance chemotherapy using S-1(MC-S1) in patients with N3 stage nasopharyngeal carcinoma achieved superior survival. The MC-S1 was administered for at least 12 cycles. The toxicities of MC-S1 were mild and tolerable.

However, whether or not dCCRT follow maintenance therapy with S-1 improve the survival outcomes of patients with locally advanced unresectable esophageal cancer are unclear. Therefore, the aim of this study is to evaluate the efficacy and side effects of patients with locally advanced unresectable esophageal cancer after dCCRT with platinum-based chemotherapy follow maintenance therapy with S-1. The primary endpoint is overall survival (OS) rates at 24 months, defined as the proportion of patients who have not experienced death from any cause at months. With a sample size of 60 patients, the study had a power of 80%, assuming 2-year OS of 45% in the experimental arm and 30% in the historical control, with a one-sided significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

1. an age of at least 20 years;
2. patients with histologically confirmed diagnosis of ESCC (Esophageal squamous cell carcinoma), GEJC (gastroesophageal junction cancer), EAC (Esophageal adenocarcinoma)
3. stage II-IVA, AJCC, 8th, locally advanced disease is suitable for dCCRT and is ineligible for curative surgery (including those who are unable or unwilling to undergo surgery)
4. an Eastern Cooperative Oncology Group performance-status score of 0-1
5. definitive concurrent chemoradiotherapy according to regional oncology guidelines for esophageal cancer, with the following criteria:

   * patients must have received platinum-based chemotherapy (at least 2 cycles of tri-weekly regimen or at least 4 cycles of weekly regimen) and radiation therapy consistent with definitive treatment (50-64 Gy)
   * no evidence of radiographic disease progression per RECIST v1.1, as documented by comparison of scans (pre- and post-definitive concurrent chemoradiotherapy) prior to enrollment.
6. adequate bone marrow, hepatic, renal and cardiac function

Exclusion Criteria:

1. patients had distant metastasis
2. patients had esophageal perforation or esophageal fistula
3. patients had tumor bleeding
4. patients had severe infection
5. History of malignancy other than esophageal cancer within 2 years prior to screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | 24 months

IPD SHARING:
Plan to Share IPD: No